CLINICAL TRIAL: NCT01632566
Title: A Multiple-Dose, Dose-Escalation Study to Evaluate the Safety and Tolerability of LY3031207 in Healthy Subjects
Brief Title: A Multiple-dose Study of LY3031207 in Healthy Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Elevation of alanine aminotransferase (ALT) and aspartate aminotransferase (AST) in some participants.
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14284; I5W-EW-LBCB (Other: Eli Lilly and Company)
Record Dates: First submitted 2012-06-25; First posted 2012-07-03 (Estimated); Results first posted 2019-06-27 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-03

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — LY3031207; Celecoxib; Simvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Daily oral administration of placebo for 28 days. Dose will match corresponding LY3031207 dosage.
  Interventions: Drug: Placebo
- LY3031207 (Experimental): Daily oral administration of 25 milligrams (mg) LY3031207 up to 450 mg LY3031207 for 28 days.
  Interventions: Drug: LY3031207
- Celecoxib (Active Comparator): Daily oral administration of 400 mg celecoxib for 28 days. Positive control for LY3031207.
  Interventions: Drug: Celecoxib
- LY3031207 + Simvastatin (Other): Daily oral administration of 75 mg LY3031207 or 225 mg LY3031207 for 28 days. Single, oral 10 mg simvastatin open-label dose administered before and after 28-day dosing of LY3031207.
  Interventions: Drug: Simvastatin

INTERVENTIONS:
Drug: Placebo — Capsules administered orally
  Arms: Placebo
Drug: LY3031207 — Administered orally
  Arms: LY3031207
Drug: Celecoxib — Administered orally
  Arms: Celecoxib
Drug: Simvastatin — Administered orally
  Arms: LY3031207 + Simvastatin

SUMMARY:
The purposes of this study are to look at safety, how well the study drug is tolerated, how much of the study drug gets into the blood stream, and how long it takes the body to get rid of it when given to healthy Japanese and non-Japanese participants as multiple doses. In addition, effects of 28-day oral dosing of LY3031207 on the amount of a cholesterol-lowering drug (simvastatin) that gets into the blood stream and how long the body takes to get rid of it will be determined. The effects of LY3031207 after single and 28-day dosing on blood pressure will also be studied. Information about any side effects that may occur will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Overtly healthy individuals based on the history and physical examinations as determined by the investigator, including first generation Japanese
* Body mass index between 17.0 and 32.0 kilograms per square meter (kg/m^2), inclusive

Exclusion Criteria:

* Have known allergies to LY3031207 or any components of the formulation, simvastatin or related compounds (other 3-Hydroxy-3-Methyl-Glutaryl-CoA [HMG CoA] reductase inhibitors), celecoxib, or sulfonamides. Participants with known aspirin allergy or allergic reaction to nonsteroidal anti-inflammatory drugs (NSAIDs) should also be excluded

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri, 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Honolulu, Hawaii, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Study enrolled participants of both Japanese and non-Japanese decent. Participants were pooled regardless of ethnicity. Participants assigned to 75 milligrams (mg) LY3031207 and 225 mg LY3031207 underwent identical procedures as those assigned to 25 mg LY3031207 with the addition of 10 mg open-label simvastatin administration on Days -3 and 28.
Groups:
- 25 mg LY3031207: Daily oral administration of 25 milligrams (mg) LY3031207 for 28 days.
- 75 mg LY3031207 and Simvastatin: Daily oral administration of 75 mg LY3031207 for up to 28 days. In addition, participants received oral administration of 10 mg open-label simvastatin on Days -3 and 28.
- 225 mg LY3031207 and Simvastatin: Daily oral administration of 225 mg LY3031207 for up to 22 days. In addition, participants received oral administration of 10 mg open-label simvastatin on Day -3 only.
- Placebo With or Without Simvastatin: Daily oral administration of placebo for up to 28 days with or without oral administration of 10 mg open-label simvastatin on Days -3 and 28.
- 400 mg Celecoxib With or Without Simvastatin: Daily oral administration of 400 mg celecoxib for up to 28 days with or without oral administration of 10 mg open-label simvastatin on Days -3 and 28.
Period: Overall Study
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin | Placebo With or Without Simvastatin | 400 mg Celecoxib With or Without Simvastatin
Started | 8 | 10 | 9 | 6 | 6
Received at Least One Dose LY3031207 | 8 | 10 | 9 | 0 | 0
Received at Least One Dose Simvastatin | 0 | 10 | 9 | 4 | 4
Completed | 8 | 7 | 0 | 4 | 4
Not Completed | 0 | 3 | 9 | 2 | 2
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Sponsor Decision | 0 | 2 | 9 | 2 | 2

BASELINE CHARACTERISTICS:
Population: Participants who received at least dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin | Placebo With or Without Simvastatin | 400 mg Celecoxib With or Without Simvastatin | Total
Number analyzed (Participants) | 8 | 10 | 9 | 6 | 6 | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (11.8) | 39.0 (11.5) | 45.1 (14.7) | 52.7 (5.8) | 44.0 (7.8) | 43.0 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 4 | 2 | 0 | 9
  Male | 7 | 8 | 5 | 4 | 6 | 30
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 0 | 0 | 0 | 1
  Not Hispanic or Latino | 7 | 10 | 9 | 6 | 6 | 38
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 3 | 3 | 2 | 12
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 5 | 6 | 3 | 2 | 4 | 20
  More than one race | 1 | 2 | 3 | 1 | 0 | 7
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 10 | 9 | 6 | 6 | 39

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug Related Adverse Events (AEs) or Any Serious AEs
Description: A treatment emergent adverse event (TEAE) is defined as an adverse event (AE) that occurs postdose or that is present predose and becomes more severe postdose. AEs presented are of all causalities and all severities.
  A summary of serious and other non-serious AEs regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline to study completion (treatment completion and follow-up, up to 35 weeks)
Population: Participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Groups:
- 10 mg Simvastatin: Oral administration of 10 mg open-label simvastatin on Days -3 and 28 for participants randomized to 75 mg LY3031207, 225 mg LY3031207 (Day -3 only), placebo, or celecoxib. Adverse events occurring following simvastatin dosing on Day -3 but prior to study drug dosing on Day 1 were counted under simvastatin.
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin | Placebo With or Without Simvastatin | 400 mg Celecoxib With or Without Simvastatin | 10 mg Simvastatin
Number analyzed (Participants) | 8 | 10 | 9 | 6 | 6 | 27
Participants
  Participants with one or more AEs | 3 | 5 | 9 | 1 | 1 | 3
  Participants with one or more serious AEs | 0 | 0 | 2 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of LY3031207
Description: Maximum concentration (Cmax) of LY3031207 post-repeated once daily doses at Day 28. Day 28 results were not calculated for participants who received 225 mg LY3031207 because the study was terminated prior to participants reaching 28 days of dosing for this treatment arm.
Time Frame: Predose up to 48 hours post last dose at Day 28
Population: Participants who received at least one dose of LY3031207 with evaluable Cmax data at Day 28. Participants who had incomplete data due to early discontinuation were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin
Number analyzed (Participants) | 8 | 6 | 0
nanograms/milliliter (ng/mL) | 1120 (34.3) | 2290 (42.4) |

3. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3031207
Description: Area under the concentration versus time curve in a dosing interval (AUC[0-tau]) of LY3031207 post-repeated once daily doses at Day 28. Day 28 results were not calculated for participants who received 225 mg LY3031207 because the study was terminated prior to participants reaching 28 days of dosing for this treatment arm.
Time Frame: Predose up to 48 hours post last dose at Day 28
Population: Participants who received at least one dose of LY3031207 with evaluable AUC (0-tau) data at Day 28. Participants who had incomplete data due to early discontinuation were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (hr*ng/mL)
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin
Number analyzed (Participants) | 8 | 6 | 0
nanograms*hours/milliliter (hr*ng/mL) | 12000 (39.7) | 30400 (45.0) |

4. Secondary Outcome: Pharmacokinetics: Time of Maximum Concentration (Tmax) of LY3031207
Description: Time of maximum concentration (Tmax) of LY3031207 post-repeated once daily doses at Day 28. Day 28 results were not calculated for participants who received 225 mg LY3031207 because the study was terminated prior to participants reaching 28 days of dosing for this treatment arm.
Time Frame: Predose up to 48 hours post last dose at Day 28
Population: Participants who received at least one dose of LY3031207 with evaluable Tmax data at Day 28. Participants who had incomplete data due to early discontinuation were not analyzed.
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin
Number analyzed (Participants) | 8 | 6 | 0
hours | 2.00 [1.02 to 4.00] | 3.00 [2.00 to 12.0] |

5. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax) of Simvastatin
Time Frame: Predose up to 48 hours post dose at Day -3 and Day 28
Population: Participants dosed with 75 mg LY3031207 from Days 1 through 28 and with oral administration of 10 mg open-label simvastatin on Days -3 and 28 and who had complete pharmacokinetic profiles following both simvastatin dosing events. Participants who had incomplete data due to early discontinuation were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms/milliliter (ng/mL)
Groups:
- 10 mg Simvastatin Day -3: Oral administration of 10 mg open-label simvastatin on Day -3 for participants randomized to 75 mg LY3031207, 225 mg LY3031207, placebo, or celecoxib.
- 10 mg Simvastatin Day 28: Oral administration of 10 mg open-label simvastatin on Day 28 for participants randomized to 75 mg LY3031207, 225 mg LY3031207, placebo, or celecoxib.
Arm/Group | 10 mg Simvastatin Day -3 | 10 mg Simvastatin Day 28
Number analyzed (Participants) | 5 | 5
nanograms/milliliter (ng/mL) | 1.78 (55.3) | 3.4 (69.3)

6. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of Simvastatin
Description: Area under the concentration versus time curve over the range of all measureable concentrations (AUC[0-tlast]) of simvastatin.
Time Frame: Predose up to 48 hours post dose at Day -3 and Day 28
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hours/milliliter (hr*ng/mL)
Arm/Group | 10 mg Simvastatin Day -3 | 10 mg Simvastatin Day 28
Number analyzed (Participants) | 5 | 5
nanograms*hours/milliliter (hr*ng/mL) | 5.23 (48.9) | 8.97 (70.1)

7. Secondary Outcome: Pharmacokinetics: Time of Maximum Concentration (Tmax) of Simvastatin
Time Frame: Predose up to 48 hours post dose at Day -3 and Day 28
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | 10 mg Simvastatin Day -3 | 10 mg Simvastatin Day 28
Number analyzed (Participants) | 5 | 5
hours | 2.00 [1.00 to 2.00] | 1.15 [1.08 to 2.00]

8. Secondary Outcome: Change From Baseline to Day 28 in Urinary Prostacyclin I (PGI) Metabolite Excretion
Time Frame: Baseline, Predose up to 12 hours prior to last dose at Day 28
Population: Zero participants were analyzed. Data not collected.
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline to Day 28 in Urinary Prostaglandin E (PGE) Metabolite Excretion
Time Frame: Baseline, Predose up to time of last dose at Day 28
Population: Zero participants were analyzed. Data not collected.
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin
Number analyzed (Participants) | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline to Day 28 in Urinary Thromboxane A (TXA) Metabolite Excretion
Time Frame: Baseline, Predose up to 12 hours prior to last dose at Day 28
Population: Zero participants were analyzed. Data not collected.
Arm/Group | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Placebo With or Without Simvastatin | 25 mg LY3031207 | 75 mg LY3031207 and Simvastatin | 225 mg LY3031207 and Simvastatin | 400 mg Celecoxib With or Without Simvastatin | 10 mg Simvastatin
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/8 | 0/10 | 2/9 | 0/6 | 0/27
Other Adverse Events (participants affected / at risk) | 1/6 | 3/8 | 5/10 | 9/9 | 1/6 | 3/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo With or Without Simvastatin (N=6) | 25 mg LY3031207 (N=8) | 75 mg LY3031207 and Simvastatin (N=10) | 225 mg LY3031207 and Simvastatin (N=9) | 400 mg Celecoxib With or Without Simvastatin (N=6) | 10 mg Simvastatin (N=27)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo With or Without Simvastatin (N=6) | 25 mg LY3031207 (N=8) | 75 mg LY3031207 and Simvastatin (N=10) | 225 mg LY3031207 and Simvastatin (N=9) | 400 mg Celecoxib With or Without Simvastatin (N=6) | 10 mg Simvastatin (N=27)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0)
Sensitivity of teeth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Irritability (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced liver injury (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Laceration (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1) | 4 (5) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Lilly voluntarily discontinued dosing of LY3031207 for all participants in LBCB because of early discontinuation criteria being met. Data for some endpoints (including blood pressure and Japanese comparison) were incomplete for the planned analyses.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days